CLINICAL TRIAL: NCT06059352
Title: Contribution of Central Auditory Processing Disorder (CAPD) to Sleep Disturbances in Autism Spectrum Disorder (ASD)
Brief Title: Sleep and Central Auditory Processing Disorder in Autism Spectrum Disorder
Acronym: ASD
Status: Recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Sponsor
Other Study IDs: 5210160
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Central Auditory Processing Disorder; Autism Spectrum Disorder; Sleep Disturbance
MeSH Terms: conditions — Language Development Disorders; Autism Spectrum Disorder; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD+ CAPD: This group includes children and adolescence with ASD who also have CAPD. No intervention will be applied to this group.
- ASD- CAPD: This group includes children and adolescence with ASD who are not affected by CAPD. No intervention will be applied to this group.

SUMMARY:
The proposed study aims to understand poor sleep as a possible cause to CAPD in children and adolescents with ASD (ASD+) compared to ASD youth without CAPD (ASD-), using both caregiver-report and objective clinician administered measures. Additionally, the study will aim to understand the complex relationship between CAPD, sleep, and other associated phenotypic features of ASD such as executive and psychiatric functioning.

DETAILED DESCRIPTION:
Participation will involve one assessment session approximating 4 hours including administration of neurocognitive and socioemotional measures by trained research staff. The research team then will determine which participants meet CAPD diagnostic criteria for both the SCAN-3 and RGDT tests and assign them to the ASD+ group. Participants not meeting these criteria will be assigned to the ASD- group. Following the assessment visit, all participants will then be asked to wear actigraphy monitors (comparable to overnight polysomnography) regularly for 14 days during nighttime sleep to objectively measure sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosis of Autism Spectrum Disorder confirmed by the Autism Diagnostic Observation Schedule and the Social Communication Questionnaire, Lifetime Version which will be filled by the parent
* IQ of 50 or higher on the Abbreviated Battery IQ Score

Exclusion Criteria:

* No confirmed diagnosis of Autism Spectrum Disorder
* History of sleep apnea
* History of restless leg syndrome
* History of any neurological disorders (e.g., seizures, tumors, etc.)
* Significant substance use in the past six months
* Inpatient hospitalization in the past three months-period

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: One hundred school-aged children and adolescents with ASD who are between the ages of 6-17 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensory Processing Patterns in Children Ages 14 and Below | Through study completion, an average of one year
  Sensory sensitivity is a composite measurement using the 86 item Sensory Profile 2 (SP-2). SP-2 has 4 quadrants; Seeking (degree child obtains sensory input); Avoiding (degree child is bothered by sensory input); Sensitivity ( degree child detects sensory input); Registration (degree child misses sensory input). SP-2 is completed by parents of subjects using a scale of 5 (almost always = 90% or more), 4 (frequently= 75% of the time), 3 (half of the time = 50%), 2 (occasionally= 25%), 1 (almost never = 10% or less), or does not apply.
  Seeking quadrant normal limits are 20-47; elevated seeking scores are ≥ 48, reduced seeking behaviors are ≤ 19.
  Avoiding quadrant normal limits are 21-46; elevated avoiding scores are ≥ 47; reduced avoiding scores are ≤ 20.
  Sensitivity quadrant normal limits are 18- 42; elevated scores are ≥ 43; reduced scores are ≤ 17 and below. Registration quadrant normal limits are 19-43; elevated scores are ≥ 44; reduced scores are ≤18.
Sensory Processing Patterns in Children Ages 15 and Above | Through study completion, an average of one year
  Sensory sensitivity is a composite measurement using the 60-item adolescent/ adult sensory profile (AASP). AASP has 4 quadrants: Low Registration, Sensation Seeking, Sensitivity; Avoiding. Subjects will respond using a scale of almost never (5% or less of the time), seldom (25% of the time), occasionally (50% of the time), frequently (75% of the time), and almost always (95% or more of the time).
  Low Registration normal limits are 27-40; elevated scores are ≥ 41; reduced registration scores are ≤ 26.
  Sensation seeking normal limits are 42-58; elevated sensation scores are ≥ 59; reduced sensation scores are ≤ 25.
  Sensitivity normal limits are 26-40; elevated sensitivity scores are ≥ 41; reduced scores are ≤ 25.
  Avoiding normal limits are 26-40; elevated scores are ≥ 41; reduced scores are ≤ 25.

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Nair, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No